CLINICAL TRIAL: NCT05215548
Title: A Phase II Study of Primary Tumor Resection for Stage IV Non-small-cell Lung Cancer Without Progression After First-line Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor
Brief Title: Primary Tumor Resection With EGFR TKI for Stage IV NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202107141RINB
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: NSCLC Stage IV
Keywords: epidermal growth factor receptor tyrosine inhibitor; lung adenocarcinoma; surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I : Surgery group (Experimental): The surgery group would receive take 12 weeks of EGFR TKI before randomization. After randomization, the surgery group would receive thoracic surgery with maximal regional control intent. Patients continue afatinib 1 to 2 weeks after surgery until disease progression or unacceptable toxicity. The residual local and metastatic sites of disease could undergo either surveillance or maintenance radio-treatment at the discretion of the treating physician.
  Interventions: Procedure: therapeutic thoracic surgery; Drug: Afatinib
- Group II : Maintenance group (Active Comparator): The control group would receive take 12 weeks of EGFR TKI before randomization. After randomization, the control group would receive afatinib until disease progression or unacceptable toxicity. The residual local and metastatic sites of disease could undergo either surveillance or maintenance radio-treatment at the discretion of the treating physician.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Procedure: therapeutic thoracic surgery — The surgery group would receive therapeutic thoracic surgery with maximal local regional control intent and would prescribe with maintenance afatinib therapy after operation. Patients continue afatinib 1 to 2 weeks after surgery.
  Arms: Group I : Surgery group
Drug: Afatinib — The patient take afatinib treatment for 12 weeks treatment and then receive systemic image study examination before randomization. If exam result showed progression the patient would be excluded from the study. Treatment response was evaluated according to the Response Evaluation Criteria in Solid Tumors (version 1.1).
  Other Names: Giotrif; BIBW 2992

SUMMARY:
Our project is going to enroll patients with stage IV NSCLC with EGFR mutation and evaluate whether primary tumor resection after receiving the afatinib can prolong survival. This project is supposed to establish a new treatment protocol for stage IV NSCLC with EGFR mutation.

DETAILED DESCRIPTION:
In Taiwan, non-small cell lung cancer (NSCLC) has been the leading cause of cancer death, making a phenomenal impact on public health. By understanding the oncogenic driver mutations of NSCLC (e.g. EGFR mutation or ALK rearrangement), the target therapy has taken the place of chemotherapy for its effectiveness and specificity, becoming the new standard of care for stage IV NSCLC. Despite the progress of medical treatment, the majority of patients with stage IV NSCLC still underwent disease progression after a period of time. Noticeably, more than half of the progression was restricted to the original sites of the tumor. It brings up the hypothesis that a combination of local consolidative therapy (e.g. surgery or radial therapy) and medical treatment could be beneficial for these patients. This has been advocated by the latest clinical trials as well.

Our project is going to enroll patients with stage IV NSCLC with EGFR mutation and evaluate whether primary tumor resection after receiving the afatinib can prolong the progression-free survival. This project is supposed to establish a new treatment protocol for stage IV NSCLC with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Stage IV non-small cell lung cancer which is amenable to thoracic surgery
* Patients must have one of the following:NSCLC which harbors EGFR exon 19 deletion or L858R mutation.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Candidate for therapeutic intent surgery to at least one site of disease
* Signed and dated written informed consent prior to admission to the study in accordance with International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use (ICH)-Good Clinical Practice (GCP) guidelines and to the local legislation

Exclusion Criteria:

* Life expectancy <= 12 weeks
* With underlying diseases such as moderate to severe Chronic Obstructive Pulmonary Disease or tuberculosis
* With uncontrol diseases including acute infection, unstable angina or angina in recent 3 months, Heart failure(NYHA≥2), myocardial infarction in recent 6 months, severe arrhythmia, moderate to severe cirrhosis, moderate to severe chronic renal insufficiency, immune insufficiency, any systemic disease with poor prognosis after treatment.
* With Cerebrovascular Accident complicated dependent activities of daily living.
* Any other cancer with active treatment in recent 5 years.
* receive thoracic surgery in the ipsilateral site with the lung cancer previously. （the biopsy surgery required for the diagnosis of lung cancer was not excluded)
* pregnant or breast-feeding woman
* Previous treatment with other EGFR TKI. NOTE: Patients who are receiving initial afatinib (6-12 weeks) outside this study are not excluded
* Disagree to receive Next Generation Sequencing for the lesion specimen after surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
2 year progression free survival rate | start date of afatinib assessed up to 2 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.

SECONDARY OUTCOMES:
Progression free survival | From the start date of afatinib assessed up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
Overall survival | From the start date of afatinib assessed up to 4 years
  Will be estimated using Kaplan-Meier method. The stratified log-rank test will be performed to test the difference in time-to-event distributions between treatment groups. Stratified Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis and to estimate hazard ratios.
Treatment-related adverse events | From the start date of afatinib assessed up to 4 years
  It refers to the number of adverse events related to afatinib monotherapy or platinum-based chemotherapy as evaluated according to CTCAE v4.0.
R0 resection rate | From the start date of afatinib assessed up to 12 weeks
  It is defined as the proportion of patients with negative surgical margin and no residual found under microscope after resection in all patients who have completed the thoracic surgery treatment.
resistant mutation events | 12 weeks to 4 years
  Patient in the surgery and control group would receive next generation sequencing for tumor mutation check. The surgery group would receive next generation sequencing twice (1. after surgery 2. progression of disease or unacceptable toxicity.) The control group would receive next generation sequencing once (progression of disease or unacceptable toxicity.)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei